CLINICAL TRIAL: NCT06239532
Title: A Single-arm, Prospective Study of HAIC Sequential TAE Combined With Tislelizumab and Surufatinib in Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: HAIC Sequential TAE Combined With Tislelizumab and Surufatinib in Unresectable Intrahepatic Cholangiocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Principal Investigator, Zhang Zongli, Professor, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REACH-01
Record Dates: First submitted 2023-12-28; First posted 2024-02-02 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — tislelizumab; surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAE+HAIC+Tislelizumab+Surufatinib (Experimental): Patients will receive hepatic arterial infusion chemotherapy (HAIC) sequential transcatheter arterial embolization(TAE) combined with Tislelizumab and Surufatinib
  Interventions: Drug: HAIC+TAE; Drug: Tislelizumab; Drug: Surufatinib

INTERVENTIONS:
Drug: HAIC+TAE — Procedure: HAIC+TAE After successful percutaneous hepatic artery cannulation for continuous pumping of drugs. Oxaliplatin(85 mg/m2); Raltitrexed (3 mg/m2) ，continuous infusion for 3 hours. HAIC was performed at an interval of at least 21 days.
Drug: Tislelizumab — Drug: Tislelizumab(200 mg) will be administered by IV infusion every 3 weeks
Drug: Surufatinib — Drug: Surufatinib was taken orally after meals, once a day, with 3-5 capsules (50mg/capsule) each time.

SUMMARY:
This is a single center, single arm, phase II, prospective study to evaluate the safety and effectiveness of HAIC combined with TAE plus an ICI and an TKI in adult patients (aged ≥18 years) with unresectable intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
Compared with systemic intravenous chemotherapy, hepatic arterial infusion chemotherapy(HAIC) has the advantages of increasing local drug concentration and reducing systemic toxic and side effects. All patients were treated with HAIC (Oxaliplatin and Raltitrexed ). Surufatinib was taken orally after meals, once a day, with 3-5 capsules (50mg/capsule) each time； Tislelizumab was given 200mg every 3 weeks. The treatment continued until the patient developed the disease or met the other criteria for terminating the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for the trial.
2. Aged ≥18 years.
3. Histologically confirmed intrahepatic cholangiocarcinoma.
4. No other previous systematic treatment for BTC.
5. At least one measurable lesion (RECIST 1.1).
6. Eastern Cooperative Oncology Group performance status 0 or 1.
7. Life expectancy of 3 months or greater.
8. Child-Pugh classification score ≤7.

Exclusion Criteria:

1. Recurrent patients.
2. Eastern Cooperative Oncology Group performance status ≥ 2.
3. Life expectancy of less than 3 months.
4. Child-Pugh classification score > 8.
5. History of hepatic encephalopathy or liver transplantation.
6. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
7. Symptomatic pleural effusion, ascites, and pericardial effusion that require drainage.
8. Portal vein tumor thrombus (PVTT) involves both the main trunk and contralateral branch or upper mesenteric vein. Inferior vena cava tumor thrombus.
9. Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-CTLA4, etc.).
10. History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
11. The researcher considers it inappropriate to enter this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  the sum of complete response rate and partial response rate

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  Time from randomization to disease progression
Conversion to surgical resection rate | 3 months
  Defined as the proportion of patients who were successfully converted to radical resection with negative hepatic margins after the study treatment regimen was calculated
Overall survival (OS) | 24 months
  Time from randomization to death for any cause
1-year overall survival rate | 12 months
  one year overall survival rate
Disease Control rate (DCR) | 24 months
  the sum of complete response rate, partial response rate and stable disease rate
Incidence rate of adverse events | 24 months
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Zongli Zhang, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li KS, Liu Y, Zhang TZ, Xu YF, Zhang ZL. Protocol of REACH-01: a single-arm, open label, prospective study of HAIC sequential TAE combined with tislelizumab and surufatinib in unresectable intrahepatic cholangiocarcinoma. Front Pharmacol. 2024 Nov 18;15:1435639. doi: 10.3389/fphar.2024.1435639. eCollection 2024. PMID 39624833